CLINICAL TRIAL: NCT04831710
Title: Safety and Efficacy of Sintilimab(S) in Combination With Histone Deacetylase Inhibitor (Chidamide, C) in Refractory and Relapsed (R) Angioimmunoblastic T-cell Lymphoma (AT): A Single-arm, Multicenter Phase II Study(SCRAT)
Brief Title: Sintilimab in Combination With Chidamide in Refractory and Relapsed AITL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huiqiang Huang, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRAT
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Angioimmunoblastic T-cell Lymphoma
Keywords: Sintilimab; Chidamide
MeSH Terms: conditions — Immunoblastic Lymphadenopathy | interventions — sintilimab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab+Chidamide (Experimental): Participants will receive Sintilimab,200mg, ivd, d1; Chidamide,30mg,po,biw,d1-21; repeated every 3 weeks(up to 1 year) until disease progression, intolerable toxicity, death, or termination of the study for any reason.
  Interventions: Drug: Sintilimab; Drug: Chidamide

INTERVENTIONS:
Drug: Sintilimab — Sintilimab,200mg, ivd, d1
  Other Names: Tyvyt®
Drug: Chidamide — Chidamide,30mg,po,biw,d1-21
  Other Names: Epidaza

SUMMARY:
Angioimmunoblastic T-cell lymphoma (AITL) belongs to a subtype of peripheral T-cell lymphoma (PTCL) and is also a distinct type of non-Hodgkin lymphoma (NHL). The clinical outcomes of AITL is poor and optimal treatment strategies for AITL have not been fully defined. Patients with disseminated or relapsed disease have a very poor outcome, and there is no standard management for relapsed or refractory disease. Epigenetic drugs have been widely used to treat patients with refractory/relapse AITL. Several phase II clinical trails demonstrated the ORR of 33-50% in patients with r/r AITL treated with HDAC inhibitors (including Belimastat, Romidepsin, Chidamide). HDAC inhibitors are important drugs for the current treatment of AITL, but still more than half of the patients can not benefit from it. PD1/PD-L1 blockade was a potent strategy for r/r PTCL in two small sample studies. Current studies have found that HDACi can upregulate the expression of PDL1, In vivo testing of C57BL/6 mice revealed a synergistic tumor suppression after combining HDACi and PD-1 blockade. We carried out a single, open-label, multicenter clinical trial enrolled patients with relapsed/refractory AITL to investigate the safety and efficacy of sintilimab in combination with chidamide.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research; fully understand and know the research and sign the Informed Consent Form (ICF); willing to follow and have the ability to complete all trial procedures;
2. Aged 18-75 years old male or female;
3. Angioimmunoblastic T-cell lymphoma confirmed by histopathology examination;
4. Paraffin tissue specimens or fresh puncture tissue specimens are available;
5. Patients with refractory or relapsed angioimmunoblastic T-cell lymphoma after anthracycline-contained regimen treatment. Refractory is defined as: patients did not get partial remission (PR) or better responses after first line treatment or disease progression within 6 months of the last protocol;
6. Eastern cooperative oncology group score: 0-1;
7. Estimated survival ≥ 3 months;
8. There must be at least one evaluate able or measurable lesion that meets the RECIL 2017 Lymphoma criteria [evaluable lesion: 18Ffluorodeoxyglucose/ Positron Emission Tomography (18FDG/PET) examination showing increased lymph node or extranodal uptake (higher than liver) and PET and/or computed tomography (Computed Tomography) CT) features are consistent with lymphoma findings; lesions can be measured: nodular lesions > 15mm or extranodal lesions > 10mm (if the only measurable lesion has received radiotherapy in the past, there must be evidence of radiological progress after radiotherapy), and accompanied by increased 18FDG uptake). Except for this, there is no measurable increase in diffuse 18FDG uptake in the liver;
9. Adequate organ and bone marrow function, no severe hematopoietic dysfunction, cardiac, pulmonary, liver, kidney, thyroid dysfunction and immune deficiency (no blood transfusion, granulocyte colony stimulating factor or other medical support was received within 14 days prior to the use of the research drug): 1) The absolute value of neutrophils (>1.0×10^9/L); 2) platelet count (> 75×10^9/L); 3) Hemoglobin (> 9 g/ dL); 4) Upper Limit Normal (ULN) or creatinine clearance rate (>40 mL/ min) of serum creatinine (<1.5 times normal value upper limit) (estimated by Cockcroft-Gault formula); 5) Serum total bilirubin < 1.5 times ULN; 6) Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) = 2.5 times ULN; 7) Coagulation function: International Normalized Ratio (INR) = 1.5 times ULN; Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) = 1.5 times ULN (unless the subject is receiving anticoagulant therapy and PT and APTT are using anticoagulant therapy at screening time). Within the expected range; 8) Thyrotropin (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) were all within the normal range (+10%);
10. There was no evidence that subjects had difficulty breathing at rest, and the measured value of pulse oximetry at rest was more than 92%;
11. Participants must pass a pulmonary function test (PFT) to confirm that forced expiratory volume (FEV1)/forced vital capacity (FVC) in the first second is more than 60%, unless it is a large mediastinal mass caused by lymphoma that cannot meet this standard; carbon monoxide diffusion (DLCO), FEV1 and FVC are all above 50% of the predicted value; all PFT results must be obtained within four weeks before the first administration;
12. Subjects who have received antineoplastic therapy should be admitted to the group only after the toxicity of the previous treatment has returned to the level of Common Terminology Criteria for Adverse Events (CTCAE) V5.0 grade score < 1 or baseline level; the level 2 toxicity caused by previous antineoplastic treatment is irreversible and is not expected to deteriorate during the study period. (e.g. thrombocytopenia, anemia, neurotoxicity, alopecia and hearing loss) can be enrolled with the consent of the researchers;
13. Women of Childbearing Potential (WOBCP) must undergo a serum pregnancy test within seven days before the first medication and the results are negative. WOBCP or men and their WOBCP partners should agree to take effective contraceptive measures from the signing of ICF until six months after the last dose of the research drug is used.

Exclusion Criteria:

1. Hemophagocytic syndrome;
2. Primary central nervous system lymphoma or secondary central nervous system involvement;
3. Received organ transplantation in the past;
4. Patients who received allogeneic hematopoietic stem cell transplantation within three years before the drug was given (patients who received allogeneic hematopoietic stem cell transplantation more than three years before the drug was given and who currently have no graft-versus-host response can be enrolled);
5. Participating in other clinical studies or planning to start this study is less than 4 weeks from the end of the previous clinical study;
6. Autologous hematopoietic stem cell transplantation was performed within 90 days before the start of the study;
7. Treated with immune checkpoint inhibitors or histone deacetylase inhibitors within one year before administration;
8. Patients with active autoimmune diseases requiring systematic treatment in the past two years (hormone replacement therapy is not considered systematic treatment, such as type I diabetes mellitus, hypothyroidism requiring only thyroxine replacement therapy, adrenocortical dysfunction or pituitary dysfunction requiring only physiological doses of glucocorticoid replacement therapy); Patients with autoimmune diseases who do not require systematic treatment within two years can be enrolled;
9. Begin the study on subjects requiring systemic glucocorticoid therapy or other immunosuppressive therapy for a given condition within 14 days before treatment [allowing subjects to use local, ocular, intra-articular, intranasal and inhaled glucocorticoid therapy (with very low systemic absorption); and allowing short-term (< 7 days) glucocorticoid prophylaxis (e.g., contrast agent overdose) Sensitivity) or for the treatment of non-autoimmune diseases (e.g. delayed hypersensitivity caused by contact allergens);
10. In the past five years, patients with other malignant tumors have undergone radical treatment, except for basal cell carcinoma of skin, squamous cell carcinoma of skin, carcinoma in situ of breast and carcinoma in situ of cervix.
11. Begin the study and receive systemic antineoplastic therapy within 28 days before treatment, including chemotherapy, immunotherapy, biotherapy (cancer vaccine, cytokines, or growth factors that control cancer), etc.;
12. The study began with major surgery within 28 days before treatment or radiotherapy within 90 days before treatment;
13. Start the study and receive Chinese herbal medicine or Chinese patent medicine treatment within 7 days before treatment;
14. Begin research on live vaccination (except influenza attenuated vaccine) within 28 days before treatment;
15. History of human immunodeficiency virus (HIV) infection and/or patients with acquired immunodeficiency syndrome are known;
16. Patients with active hepatitis B or active hepatitis C. Patients who are positive for hepatitis B Surface Antigen (HBsAg) or hepatitis C Virus (HCV) antibodies at screening stage must pass further detection of hepatitis B Virus (HBV) DNA titer (no more than 2500 copies/mL or 500 IU/mL) and HCV RNA (no more than the lower limit of the detection method) in the row. In addition to active hepatitis B or hepatitis C infections requiring treatment, group trials can be conducted. Hepatitis B carriers, stable hepatitis B (DNA titer should not be higher than 2500 copies/mL or 500 IU/mL) after drug treatment, and cured hepatitis C patients can be enrolled in the group;
17. Patients with active pulmonary tuberculosis;
18. Start studying any active infections requiring systemic anti-infective treatment within 14 days of treatment.
19. Pregnant or lactating women;
20. People with known history of alcoholism or drug abuse;
21. Have uncontrollable complications, including but not limited to symptomatic congestive heart failure, uncontrollable hypertension, unstable angina, active peptic ulcer or hemorrhagic diseases;
22. History of interstitial lung disease or non-infectious pneumonia. Subjects who had previously had non-infectious pneumonia caused by drugs or radiation but had no symptoms were allowed to enter the group;
23. The QTcF interval is more than 450 msec, unless it is secondary to bundle branch block;
24. Past psychiatric history; incapacitated or restricted;
25. According to the researchers' judgment, patients' underlying condition may increase their risk of receiving research drug treatment, or confuse their judgment on toxic reactions;
26. Other researchers consider it unsuitable for patients to participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR), complete response rate (CRR), partial response rate (PRR) | Up to 24 months
  Assessed by the RECIL 2017 Response Criteria for Malignant Lymphoma

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 24 months
  PFS is defined as the time from the treatment date to the date of disease progression per the RECIL 2017 Response Criteria for Malignant Lymphoma or death regardless of cause.
Overall Survival (OS) | Up to 24 months
  OS is defined as the time from treatment to the date of death.
Duration of Response (DOR) | Up to 24 months
  Among participants who experience an objective response, DOR is defined as the date of their first objective response (which is subsequently confirmed) to disease progression per the RECIL 2017 Response Criteria for Malignant Lymphoma or death regardless of cause.
Time to disease response (TTR) | Up to 24 months
  Among participants who experience an objective response, TTR is defined as the date of their first administration to the day of their first objective response (which is subsequently confirmed) per the RECIL 2017 Response Criteria for Malignant Lymphoma.
Time to progression (TTP) | Up to 24 months
  Among all participants, TTP is defined as the date of their first administration to the day of disease progression per the RECIL 2017 Response Criteria for Malignant Lymphoma or death regardless of cause.
The frequency of adverse events (adverse events, AEs) and serious adverse events (SAEs) | Up to 24 months
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAE were defined as AEs with onset during the treatment period or that are a consequence of a pre-existing condition that has worsened since baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China